CLINICAL TRIAL: NCT03495466
Title: Comparison of Local Only Anesthesia Versus Sedation in Patients Undergoing Bilateral Carpal Tunnel Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kanu Goyal, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015H0148
Record Dates: First submitted 2018-03-20; First posted 2018-04-12 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Bilateral Carpal Tunnel Syndrome (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local only Anesthesia (Active Comparator): The patient will receive local only anesthesia during the first surgery and local with sedation anesthesia for their second surgery.
  Interventions: Procedure: Local only anesthesia vs Local with sedation anesthesia
- Local with sedation anesthesia (Active Comparator): The patient will receive local with sedation anesthesia during the first surgery and local only anesthesia for their second surgery.
  Interventions: Procedure: Local only anesthesia vs Local with sedation anesthesia

INTERVENTIONS:
Procedure: Local only anesthesia vs Local with sedation anesthesia — The investigators are comparing two approved sedation types that are using during carpal tunnel surgery.

SUMMARY:
The study design is a prospective randomized control trial. Four surgeons will enroll up to 30 patients in the study. Patients will be asked to participate if they plan to undergo bilateral carpal tunnel release with one of the study surgeons, are greater than 18 years of age but younger than 89, have had no prior carpal tunnel surgery, and agree to undergo carpal tunnel surgery under two different types of anesthesia. If patients meet these criteria and agree to participate in the study, they will be consenting to have one hand operated on with local only anesthesia and the other hand with local anesthesia with sedation. The patient will randomly be assigned to have one of the two anesthetic methods for the first carpal tunnel release, followed by the other anesthetic for the second carpal tunnel release. The two surgeries will be completed by the same surgeon and may be performed at any time interval apart; however, the investigators will recommend that patients get the second surgery within 4 weeks of the first. The particular surgical technique of carpal tunnel release will be performed according to the individual surgeon's preference, but the same technique will be used on both wrists. The surgeon will discuss the proposed advantages and disadvantages of each anesthetic method prior to enrolling the patient (advantages and disadvantages discussed above). The treating surgeons will continue to utilize their standard surgical technique on each side, regardless of a patient's participation in the study.

ELIGIBILITY:
Inclusion Criteria:

Patients with a diagnosis of bilateral carpal tunnel syndrome and who have been recommended to undergo bilateral carpal tunnel release will be recruited to the study. Standard diagnostic criteria will be utilized by the surgeon including symptoms, objective signs on physical exam, and adjunct studies such as electromyography, nerve conduction and neuromuscular ultrasound. These patients may be identified in any of four surgeon offices, all of whom are fellowship-trained in hand and upper extremity surgery. As in standard practice, the participating surgeons will screen individuals to identify any contraindications for either method of anesthesia. Patients meeting the general inclusion and exclusion criteria listed below will be eligible to participate. Should any questions arise regarding an individual's eligibility or safety, a consultation with Dr. Mike Guertin, anesthesiologist, will be obtained. Inclusion criteria include: - Individuals who are able to give consent - Individuals who are at least 18 years of age but no older than 89. - Individuals who require bilateral carpal tunnel release surgery - Willingness to undergo each type of anesthesia

Exclusion criteria include: - Age < 18 years and > 89 years - Prior history of carpal tunnel release - Allergy to local anesthetics - Medical conditions that would exclude the participant from being a candidate for sedation during surgery (examples: respiratory conditions (chronic obstructive pulmonary disease, lung cancer, sickle cell disease); liver and kidney disease.) - Any other contraindications for sedation not listed - Unwillingness to participate in the study - Unable to consent for themselves -First surgery being performed endoscopically or open and the second surgery requiring the opposite technique - Prisoners

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Measurement of patients perspective and preferences with their surgeries (local only and local with sedation) by VAS and multiple choice questions. | measure at first post-operative appointment after each surgery, an average of 12-18 weeks
  A post-operative questionnaire has been compiled to capture study patient perspectives and preferences with their surgeries. The study patients will fill out this questionnaires during their first post-operative visits after each surgery.

SECONDARY OUTCOMES:
Measurement of individuals preferred surgery (local only and local with sedation) by VAS score | measured after both surgeries have been completed,an average of 12-18 weeks
  The study patient will be asked to rate their preferred surgery at the end of the study.
Measurement of individuals satisfaction with each surgery (local only and local with sedation) by VAS score | measured six week follow-up after each surgery
  The study patient will rate how satisfied they were after each surgery.
Measurement of level of anxiety about each type of surgery (local only and local with sedation) by Beck Anxiety Inventory (questionnaire) | measured at baseline and prior to each surgery,an average of 12-18 weeks
  Beck Anxiety Inventory will be collected at baseline and on the days of surgery to analyze any increases or decreases in anxiety.

OTHER OUTCOMES:
Cost of surgery- chart review | measured after each surgery,an average of 12-18 weeks
  The investigators will review the cost billed to the study patients insurance after each surgery.
Time in surgical facility- chart review | measured after each surgery, an average of 12-18 weeks
  The investigators will review the amount of time the study patients spent in the surgery center on the day of their surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State Wexner Medical Center, Columbus, Ohio, United States